CLINICAL TRIAL: NCT02864108
Title: Research to Develop the Human Trisome Project Biobank
Brief Title: The Human Trisome Project
Acronym: HTP
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Linda Crnic Institute for Down Syndrome (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH); GLOBAL Down Syndrome Foundation (Unknown); Anna and John J. Sie Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 15-2170; UL1TR001082 (NIH)
Record Dates: First submitted 2016-07-21; First posted 2016-08-11 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Down Syndrome; Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, mouth swab, urine (optional), stool (optional)

GROUPS / COHORTS (2):
- Those with trisomy 21: People aged 6 months to 89 years old who have some form of trisomy 21.
- Controls: People aged 6 months to 89 years old who do not have trisomy 21. These persons can be related to someone with some form of trisomy 21 but do not have to be related.

SUMMARY:
The Human Trisome Project will significantly increase the speed of Down syndrome research and the understanding of associated medical conditions. Its biobank will provide de-identified samples to research.

DETAILED DESCRIPTION:
The purpose of this study is to provide qualified and approved researchers with access to biological samples and health information to answer specific research questions. This project will significantly increase the speed of Down syndrome research and the understanding of associated medical conditions such as Alzheimer's disease, congenital heart defects, autoimmune disorders, autism, and some forms of leukemia.

Participation includes a blood draw, a mouth swab, and allowing researchers to look at your health information yearly for the next 5 years. Optional procedures include providing a urine and/or stool sample and taking part in the study for a longer time frame.

ELIGIBILITY:
Inclusion Criteria:

Anyone 6 months to 89 years old who:

1. has Down syndrome (any type)
2. does not have Down syndrome

Exclusion Criteria:

1. Prisoners
2. Wards of the state

Ages: 6 Months to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Down syndrome, individuals related to someone with Down syndrome or of the general population who do not have a relationship to Down syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-07; Primary Completion 2036-07 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants and Controls Enrolled in Biobank | 5 years
  Create biobank of blood cells and plasma, saliva, mouth swab, urine, stool, and induced pluripotent stem cells (iPSC) cells for use in approved research projects.

SECONDARY OUTCOMES:
Number of Clinical Records Available for Approved Research Purposes | 5 years
  Create a database of clinical information to pair with biological samples listed above.
Multidimensional Sample Characterization | 5 years
  Characterize biological samples with multidimensional cellular and molecular analyses to generate the most thoroughly characterized set of samples from individuals with Down syndrome in the world.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Espinosa, PhD, Principal Investigator — Linda Crnic Institute for Down Syndrome at the University of Colorado Denver
Locations (1):
- Linda Crnic Institute for Down Syndrome at the University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waugh KA, Araya P, Pandey A, Jordan KR, Smith KP, Granrath RE, Khanal S, Butcher ET, Estrada BE, Rachubinski AL, McWilliams JA, Minter R, Dimasi T, Colvin KL, Baturin D, Pham AT, Galbraith MD, Bartsch KW, Yeager ME, Porter CC, Sullivan KD, Hsieh EW, Espinosa JM. Mass Cytometry Reveals Global Immune Remodeling with Multi-lineage Hypersensitivity to Type I Interferon in Down Syndrome. Cell Rep. 2019 Nov 12;29(7):1893-1908.e4. doi: 10.1016/j.celrep.2019.10.038. PMID 31722205
- See also: The Human Trisome Project™ — http://www.trisome.org